CLINICAL TRIAL: NCT02349581
Title: Ultrasound Guided Pectoral Nerves (Pecs) Blockade in Persistent Pain After Breast Cancer Surgery
Brief Title: Ultrasound Guided Pectoral Nerves Blockade for Persistent Pain After Breast Cancer Surgery
Acronym: PPBCS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Kehlet, Henrik, M.D., Ph.D. (Individual)
Responsible Party: Principal Investigator, Nelun Wijayasinghe, Anesthesiologist, clinical researcher, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-6-2014-036
Record Dates: First submitted 2015-01-13; First posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Persistent Pain After Breast Cancer Surgery
Keywords: Anesthetics, Local; Mastectomy; Neuralgia; Nerve block
MeSH Terms: conditions — Neuralgia | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Block (Experimental): Patients with persistent pain after breast cancer surgery receive the ultrasound guided PECS block of 20mls 0.25% bupivacaine
  Interventions: Procedure: PECS block; Drug: Bupivacaine
- Sonoanatomy (No Intervention): 16 patients awaiting surgery for breast cancer were scanned using ultrasound to determine the sonoanatomy of the PECS block

INTERVENTIONS:
Procedure: PECS block — Ultrasound guided delivery of local anesthetic between the pectoral muscles
  Arms: Block
Drug: Bupivacaine
  Arms: Block

SUMMARY:
This is a pilot study of the pectoral nerves block (PECS) in patients with persistent pain after breast cancer surgery.

DETAILED DESCRIPTION:
This study is in 2 parts: Part 1 is a description of the anatomy of the PECS block in pain free, unoperated patients using ultrasonography (non invasive). Part 2 is the administration of the block to patients that have persistent pain after breast cancer surgery. Before and after the block we will take a detailed pain history and do neurophysiological tests called quantitative sensory testing (QST). These tests assess the patients' ability to feel warmth, cold and test their thresholds for pain. The block is then administered using ultrasound guidance and 20mls of 0.25% bupivacaine is injected in the pectoral muscles on the side with pain. Thirty minutes after the block, the pain is re assessed and the QST is repeated.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, aged 18 years or over, treated for breast cancer
* Patients with persistent pain in the breast after surgical treatment for breast cancer. Their pain score must be 4 or more on the numerical rating scale (NRS).

Exclusion Criteria:

* breast surgery within the last 12 months
* previous cosmetic surgery
* bilateral breast cancer (receiving bilateral intervention)
* pregnant or breast feeding
* neurological disease
* on-going treatment for severe mental illness or who abuse alcohol or drugs
* are unable to understand written or spoken Danish or English
* lack mental capacity to give informed consent or cooperate with the neurophysiological testing
* an allergy to amide local anaesthetics
* pacemaker in situ
* received treatment outside guidelines and recommendations from the Danish Breast Cancer Co-operative Group (DBCG)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Differences in summed pain intensity score (SPI) | 30 minutes after blockade
  SPI is a combination of pain at rest + pain on arm abduction + pain with 100kPa pressure. SPI will be taken before and 30 minutes after the PECS block

SECONDARY OUTCOMES:
Differences in quantitative sensory testing (QST) values | 30 minutes after blockade
  QST consists of sensory mapping (delineating areas of hypo/hyperesthesia and/or allodynia), warm detection thresholds, cool detection thresholds, heat pain thresholds, suprathermal heat pain response and pressure pain thresholds. These will be measured before and 30 minutes after the PECS block

OTHER OUTCOMES:
Longer term effects (Daily pain scores and functional questionnaire) | 1 week after blockade
  Patients will complete a pain diary for 5 consecutive days before administration of the PECS block and 7 consecutive days after the block. The patients also complete a functional questionnaire the day before the block and again exactly one week after the block.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kehlet, MD, PhD, DMsc, Study Director — Rigshospitalet, Denmark
Locations (1):
- Section for surgical pathophysiology 7621 Rigshospitalet, Copenhagen, Region Sjælland, Denmark